CLINICAL TRIAL: NCT01006122
Title: A Randomized Phase 2, Double Blind, Placebo-Controlled, Multi-Center Crossover Study Of PF-03654746 As A Daily Treatment For Excessive Daytime Sleepiness (EDS) Associated With Narcolepsy
Brief Title: A Study Of A Novel Compound For Excessive Daytime Sleepiness Associated With Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8801015
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Excessive Daytime Sleepiness; Narcolepsy
Keywords: Randomized; double-blind; placebo-controlled; crossover study of PF-03654746 in Excessive Daytime Sleepiness associated with Narcolepsy
MeSH Terms: conditions — Disorders of Excessive Somnolence; Narcolepsy | interventions — N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-03654746 (Active Comparator): At the end of the second arm of the study, the patient will have completed the study and have a 7-10 day follow-up visit.
  Interventions: Drug: PF-03654746

INTERVENTIONS:
Drug: Placebo — Patients receiving placebo will undergo the same procedures as those receiving active treatment. Each patient will receive matching placebo tablets in a fixed dose escalation schedule beginning at 0.25 mg QD for 5 days; then up to 0.50 mg QD for another 5 days; and up to 1.0 mg QD for an additional 5 days. At the end of this fixed titration schedule, the patient will either stay at 1.0 mg; decrease to 0.5 mg or increase to 2.0 mg based upon the clinicians judgment regarding efficacy and side effects at the 1.0 dose level. The patient will then remain at the determined dose for a 3 week stable dosing period, with a 7 (-2/+ 9) day wash out and then crossover to repeat the same sequence for the second arm of the study.
  Arms: Placebo
Drug: PF-03654746 — Each patient will receive PF-03654746 tablets in a fixed dose titration schedule beginning at 0.25 mg QD for 5 days; then up to 0.50 mg QD for another 5 days; and up to 1.0 mg QD for an additional 5 days. At the end of this fixed titration schedule, the patient will either stay at the 1.0 mg dose; decrease to 0.50 mg or increase to 2.0 mg based upon the clinician's judgement regarding efficacy and side effects at the 1.0 mg dose. The patient will remain at the determined dose for a 3 week stable dosing period.
  Arms: PF-03654746

SUMMARY:
Histaminergic agents are known to be involved with the sleep/wake cycle. This compound is a histaminergic agent which therefore may improve alertness and awakeness in patients with excessive daytime sleepiness (EDS) associated with narcolepsy. Significant improvement in EDS when treated with this compound compared to placebo in patients with narcolepsy is hypothesized.

ELIGIBILITY:
Inclusion Criteria:

* ISDC diagnosis of narcolepsy
* Excessive Daytime Sleepiness in association with a diagnosis of narcolepsy
* An MWT (Maintenance of Wakefulness Test) average sleep latency of under 15 minutes at Baseline

Exclusion Criteria:

* No other diagnosed sleep disorders (e.g., sleep apnea)
* Major medical disorders
* Major psychiatric disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Vernon Hills, Illinois
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Hattiesburg, Mississippi
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Dublin, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03654746 First, Then Placebo: PF-03654746 at a starting dose of 0.25 milligram (mg) to maximum dose of 2 mg, depending upon the safety and tolerability, given orally once daily as powder in a capsule (PIC) in the titration phase (TP) at 5 days interval up to 15 to 25 days, depending on dose toleration followed by a 3-week stable dose phase (SP) at fixed dose stabilized in the TP in the first double-blind (DB) intervention period then placebo matched to PF-03654746 orally once daily as PIC in the second DB intervention period. A washout period of at least 7 days was maintained between each treatment period.
- Placebo First Then, PF-03654746: Placebo matched to PF-03654746 orally once daily as PIC in the first DB intervention period then PF-03654746 at a starting dose of 0.25 mg to maximum dose of 2 mg, depending upon the safety and tolerability, given orally once daily as PIC in the TP at 5 days interval up to 15 to 25 days, depending on dose toleration followed by a 3-week SP at fixed dose stabilized in the TP in the second DB intervention. A washout period of at least 7 days was maintained between each treatment period.
Period: First Double-blind Intervention Period
Arm/Group | PF-03654746 First, Then Placebo | Placebo First Then, PF-03654746
Started | 47 | 48
Completed | 31 | 31
Not Completed | 16 | 17
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Does not meet entrance criteria | 1 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Other | 3 | 0
Not completed — Adverse Event | 0 | 4
Period: Wash-out Period (at Least 7 Days)
Arm/Group | PF-03654746 First, Then Placebo | Placebo First Then, PF-03654746
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0
Period: Second Double-blind Intervention Period
Arm/Group | PF-03654746 First, Then Placebo | Placebo First Then, PF-03654746
Started | 31 | 31
Completed | 29 | 24
Not Completed | 2 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all participants who were randomized to a treatment sequence and received at least 1 dose of study drug.
Groups:
- Entire Study: Included all participants randomized to receive PF-03654746 first and placebo first.
Arm/Group | Entire Study
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maintenance of Wakefulness Test (MWT) Score at Day 21 of Stable Dosing Phase
Description: MWT measured ability of participant to remain awake. Participants were instructed to try and remain awake during series of six 20-minute periods in a semi-recumbent position in dark room. Each period was terminated immediately after sleep onset or at end of 20 minutes if no sleep occurred. Poorest outcome was 0 minute the best was 20 minutes.
Time Frame: Baseline, Day 21 of stable dosing phase
Population: Full analysis set (FAS) consisted of all participants who were randomized to a treatment sequence and received at least 1 dose of study drug. Here "N"(number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at specified time points for each arm.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- PF-03654746: PF-03654746 at a starting dose of 0.25 milligram (mg) to maximum dose of 2 mg, depending upon the safety and tolerability, given orally once daily as powder in a capsule (PIC) in the titration phase (TP) at 5 days interval up to 15 to 25 days, depending on dose toleration followed by a 3-week stable dose phase (SP) at fixed dose stabilized in the TP in first or second DB intervention periods.
- Placebo: Placebo matched to PF-03654746 orally once daily as PIC in the first or second DB intervention periods.
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 77 | 79
minutes
  Baseline: n=77, 79 | 6.30 (4.155) | 5.81 (4.126)
  Change at Day 21 (SP): n=54, 60 | 1.29 (4.518) | 1.10 (3.878)
Statistical Analysis 1: Comparison: PF-03654746 vs Placebo; One sided p-value was based on linear mixed effects model with treatment and period as fixed effects, baseline MWT as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.418, Mixed Models Analysis; Least Squares (LS) Mean Difference = 0.16, 80% CI 2-sided [-0.81 to 1.12], Standard Error of Mean 0.747

2. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at Day 5, 10, 15, 20 of Titration Phase and Day 7, 14, 21 of Stable Dosing Phase
Description: ESS is a simple, self-administered questionnaire which provides a measurement of the participant's general level of daytime sleepiness. The participant rates the chance that he/she would fall asleep when in 8 different situations (e.g. sitting and reading, talking to someone, etc.) commonly encountered in daily life on a scale of 0 (no daytime sleep) to 3 (maximum daytime sleep). Total score was the sum of 8 situations ranges from 0 to 24 with a higher score indicating greater daytime sleepiness.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 7, 14, 21 of stable dosing phase
Population: FAS consisted of all participants who were randomized to a treatment sequence and received at least 1 dose of study drug. Here "n" signifies participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
units on a scale
  Baseline: n=78, 79 | 16.54 (4.196) | 16.32 (4.407)
  Change at Day 5 (TP): n=67, 78 | -2.06 (2.928) | -0.74 (2.770)
  Change at Day 10 (TP): n=69, 76 | -2.00 (3.325) | -1.16 (3.402)
  Change at Day 15 (TP): n=67, 74 | -2.67 (3.933) | -1.35 (4.053)
  Change at Day 20 (TP): n=59, 65 | -2.42 (3.944) | -1.74 (4.542)
  Change at Day 7 (SP): n=63, 67 | -2.92 (4.386) | -1.81 (4.743)
  Change at Day 14 (SP): n=63, 67 | -2.89 (4.618) | -1.57 (4.762)
  Change at Day 21 (SP): n=56, 61 | -2.45 (3.765) | -1.80 (5.231)
Statistical Analysis 1: Comparison: PF-03654746 vs Placebo; Day 5 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.054, Mixed Models Analysis; LS Means Difference = -0.73, 80% CI 2-sided [-1.32 to -0.15], Standard Error of Mean 0.457
Statistical Analysis 2: Comparison: PF-03654746 vs Placebo; Day 10 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.247, Mixed Models Analysis; LS Means Difference = -0.31, 80% CI 2-sided [-0.89 to 0.27], Standard Error of Mean 0.453
Statistical Analysis 3: Comparison: PF-03654746 vs Placebo; Day 15 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis; LS Means Difference = -0.60, 80% CI 2-sided [-1.19 to -0.01], Standard Error of Mean 0.457
Statistical Analysis 4: Comparison: PF-03654746 vs Placebo; Day 20 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.604, Mixed Models Analysis; LS Means Difference = 0.13, 80% CI 2-sided [-0.50 to 0.75], Standard Error of Mean 0.487
Statistical Analysis 5: Comparison: PF-03654746 vs Placebo; Day 7 (SP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.232, Mixed Models Analysis; LS Means Difference = -0.35, 80% CI 2-sided [-0.95 to 0.26], Standard Error of Mean 0.473
Statistical Analysis 6: Comparison: PF-03654746 vs Placebo; Day 14 (SP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.093, Mixed Models Analysis; LS Means Difference = -0.63, 80% CI 2-sided [-1.23 to -0.02], Standard Error of Mean 0.473
Statistical Analysis 7: Comparison: PF-03654746 vs Placebo; Day 21 (SP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline total score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.274, Mixed Models Analysis; LS Means Difference = -0.30, 80% CI 2-sided [-0.94 to 0.34], Standard Error of Mean 0.498

3. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI) Global Score at Day 5, 10, 15, 20 of Titration Phase and Day 7, 14, 21 of Stable Dosing Phase
Description: BFI is a subjective-completed tool for the assessment of the impact of fatigue on daily functioning. There are 3 questions that pertain specifically to level of fatigue and 6 questions regarding general activity level, mood and quality of life, all are answered on an 11-point scale, with "0" being "No fatigue at all" to "10" being "As bad as you can imagine". The global score is calculated by taking the sum of all 9 rating scales for a minimum score of 0 and a maximum score of 90. Higher global scores are associated with more severe fatigue.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 7, 14, 21 of stable dosing phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
units on a scale
  Baseline: n=78, 79 | 5.01 (2.564) | 5.02 (2.436)
  Change at Day 5 (TP): n=67, 78 | -1.02 (2.116) | -0.77 (1.900)
  Change at Day 10 (TP): n=68, 76 | -0.85 (1.928) | -0.88 (1.668)
  Change at Day 15 (TP): n=67, 74 | -1.18 (2.177) | -0.78 (2.193)
  Change at Day 20 (TP): n=59, 65 | -0.86 (2.104) | -0.89 (1.816)
  Change at Day 7 (SP): n=63, 67 | -0.96 (2.218) | -1.07 (2.214)
  Change at Day 14 (SP): n=63, 67 | -0.98 (2.195) | -1.11 (2.146)
  Change at Day 21 (SP): n=56, 61 | -0.74 (2.265) | -1.09 (2.248)
Statistical Analysis 1: Comparison: PF-03654746 vs Placebo; Day 5 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.121, Mixed Models Analysis; LS Means Difference = -0.29, 80% CI 2-sided [-0.60 to 0.03], Standard Error of Mean 0.244
Statistical Analysis 2: Comparison: PF-03654746 vs Placebo; Day 10 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.394, Mixed Models Analysis; LS Means Difference = -0.07, 80% CI 2-sided [-0.38 to 0.25], Standard Error of Mean 0.243
Statistical Analysis 3: Comparison: PF-03654746 vs Placebo; Day 15 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis; LS Means Difference = -0.36, 80% CI 2-sided [-0.67 to -0.04], Standard Error of Mean 0.244
Statistical Analysis 4: Comparison: PF-03654746 vs Placebo; Day 20 (TP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.495, Mixed Models Analysis; LS Means Difference = -0.00, 80% CI 2-sided [-0.34 to 0.33], Standard Error of Mean 0.260
Statistical Analysis 5: Comparison: PF-03654746 vs Placebo; Day 7 (SP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.711, Mixed Models Analysis; LS Means Difference = 0.14, 80% CI 2-sided [-0.18 to 0.46], Standard Error of Mean 0.253
Statistical Analysis 6: Comparison: PF-03654746 vs Placebo; Day 14 (SP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.767, Mixed Models Analysis; LS Means Difference = 0.18, 80% CI 2-sided [-0.14 to 0.51], Standard Error of Mean 0.253
Statistical Analysis 7: Comparison: PF-03654746 vs Placebo; Day 21 (SP), P-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects, baseline global score as a covariate and participant as random effect; Test type: Superiority or Other; p = 0.698, Mixed Models Analysis; LS Means Difference = 0.14, 80% CI 2-sided [-0.20 to 0.48], Standard Error of Mean 0.266

4. Secondary Outcome: Change From Baseline in Cataplexy Episodes at Day 7, 14, 21 of Stable Dosing Phase
Description: Cataplexy is a medical condition in which a person suffers sudden physical collapse though remaining conscious. Cataplexy episodes is number of counts the participant had cataplexy.
Time Frame: Baseline, Day 7, 14, 21 of stable dosing phase
Population: FAS consisted of all participants who were randomized to a treatment sequence and received at least 1 dose of study drug. Here "N" (number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: cataplexy episodes
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 63 | 72
cataplexy episodes
  Baseline: n=63, 72 | 5.71 (9.683) | 5.92 (12.658)
  Change at Day 7 (SP): n=53, 58 | -1.91 (6.473) | -2.67 (8.717)
  Change at Day 14 (SP): n=51, 60 | -1.71 (7.103) | -2.63 (8.471)
  Change at Day 21 (SP): n=44, 57 | -2.09 (7.882) | -2.95 (9.720)

5. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) at Day 21 of Stable Dosing Phase
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality, social functioning (SF), role emotional (RE) and mental health (MH). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Day 21 of stable dosing phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
units on a scale
  Baseline: PF (n=78, 79) | 79.68 (22.554) | 80.38 (22.882)
  Baseline: RP (n=77, 79) | 61.20 (31.305) | 65.19 (30.482)
  Baseline: BP (n=78, 79) | 68.97 (24.685) | 73.89 (26.619)
  Baseline: GH (n=78, 79) | 71.15 (16.701) | 73.03 (18.660)
  Baseline: Vitality (n=78, 79) | 38.46 (23.560) | 38.69 (21.443)
  Baseline: SF (n=78, 79) | 68.11 (28.536) | 69.30 (26.690)
  Baseline: RE (n=77, 79) | 79.65 (26.782) | 79.01 (26.550)
  Baseline: MH (n=78, 79) | 74.62 (15.411) | 77.34 (15.209)
  Change at Day 21 (SP): PF (n=55, 61) | 0.55 (15.174) | 4.75 (15.450)
  Change at Day 21 (SP): RP (n=54, 61) | 1.16 (22.191) | -1.54 (27.235)
  Change at Day 21 (SP): BP (n=55, 61) | 1.02 (16.455) | 2.23 (20.078)
  Change at Day 21 (SP): GH (n=55, 61) | -0.95 (11.762) | 0.52 (10.062)
  Change at Day 21 (SP): Vitality (n=55, 61) | 1.93 (19.833) | 1.64 (22.329)
  Change at Day 21 (SP): SF (n=55, 61) | -2.05 (18.283) | 3.48 (23.288)
  Change at Day 21 (SP): RE (n=54, 61) | -0.93 (21.577) | 6.56 (23.477)
  Change at Day 21 (SP): MH (n=55, 61) | -2.45 (11.258) | -0.25 (17.307)

6. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Scale Score
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Clinician responded to a question: "Compared to your subject's condition at the beginning of treatment, how much has your subject changed?". Improvement was compared to baseline and was defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Day 5, 10, 15, 20 of titration phase; Day 7, 14, 21 of stable dosing phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 69 | 77
units on a scale
  Day 5 (TP): n=67, 77 | 3.51 (0.859) | 3.75 (0.905)
  Day 10 (TP): n=69, 76 | 3.48 (0.994) | 3.61 (0.850)
  Day 15 (TP): n=67, 74 | 3.36 (0.980) | 3.35 (1.052)
  Day 20 (TP): n=59, 65 | 3.34 (1.124) | 3.29 (1.071)
  Day 7 (SP): n=63, 67 | 3.16 (1.139) | 3.19 (1.076)
  Day 14 (SP): n=64, 67 | 3.11 (1.210) | 3.33 (1.021)
  Day 21 (TP): n=56, 60 | 3.25 (1.210) | 3.27 (1.177)
Statistical Analysis 1: Comparison: PF-03654746 vs Placebo; Day 5 (TP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.127, Mixed Models Analysis; LS Means Difference = -0.16, 80% CI 2-sided [-0.34 to 0.02], Standard Error of Mean 0.142
Statistical Analysis 2: Comparison: PF-03654746 vs Placebo; Day 10 (TP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.303, Mixed Models Analysis; LS Means Difference = -0.07, 80% CI 2-sided [-0.25 to 0.11], Standard Error of Mean 0.141
Statistical Analysis 3: Comparison: PF-03654746 vs Placebo; Day 15 (TP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.738, Mixed Models Analysis; LS Means Difference = 0.09, 80% CI 2-sided [-0.09 to 0.27], Standard Error of Mean 0.143
Statistical Analysis 4: Comparison: PF-03654746 vs Placebo; Day 20 (TP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.850, Mixed Models Analysis; LS Means Difference = 0.16, 80% CI 2-sided [-0.04 to 0.35], Standard Error of Mean 0.152
Statistical Analysis 5: Comparison: PF-03654746 vs Placebo; Day 7 (SP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.631, Mixed Models Analysis; LS Means Difference = 0.05, 80% CI 2-sided [-0.14 to 0.24], Standard Error of Mean 0.148
Statistical Analysis 6: Comparison: PF-03654746 vs Placebo; Day 14 (SP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.160, Mixed Models Analysis; LS Means Difference = -0.15, 80% CI 2-sided [-0.34 to 0.04], Standard Error of Mean 0.147
Statistical Analysis 7: Comparison: PF-03654746 vs Placebo; Day 21 (SP), One-sided p-value was based on linear mixed effects model with treatment, period, time and treatment by time interaction as fixed effects and participant as random effect; Test type: Superiority or Other; p = 0.541, Mixed Models Analysis; LS Means Difference = 0.02, 80% CI 2-sided [-0.18 to 0.22], Standard Error of Mean 0.156

7. Other Pre Specified Outcome: Number of Participants With Vital Signs Data
Description: Criteria for potential clinical concern in vital signs: supine and standing systolic blood pressure (BP) less than (<) 90 millimeter of mercury (mmHg), supine and standing diastolic BP <50 mmHg, supine and standing heart rate <40 beats per minute (bpm) or >140 bpm. Number of participants who met the criteria for potential clinical concern was reported.
Time Frame: Baseline up to 7-10 days after Day 21 (stable dosing phase)
Population: Safety analysis set consisted of all participants who received at least 1 dose of study drug. Here "N" (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 74 | 79
participants
  Supine systolic BP: < 90 mmHg | 2 | 3
  Standing systolic BP: < 90 mmHg | 3 | 5
  Supine diastolic BP: <50 mmHg | 0 | 1

8. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory parameters included hematology (hemoglobin, hematocrit, red blood cell count, platelets, leukocytes, total neutrophils, eosinophils, basophils, lymphocytes, monocytes); liver function (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, albumin, total protein); renal function (creatinine, blood urea nitrogen, uric acid, sodium, potassium, chloride, bicarbonate, calcium); urinalysis (protein, blood), and clinical chemistry (glucose). Total number of participants with laboratory abnormalities was reported.
Time Frame: Baseline up to Day 21 of stable dosing phase
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 74 | 79
participants | 57 | 61

9. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Findings
Description: Criteria for potential clinical concern in ECG parameters: maximum PR interval of greater than or equal to (>=) 300 milliseconds (msec), maximum QRS interval >=200 msec, maximum Fridericia's correction of QT (QTcF) interval of 450 to <480 msec, 480 to <500 msec and >=500 msec. Number of participants who met the criteria for potential clinical concern in ECG findings were reported.
Time Frame: Baseline up to Day 21 of stable dosing phase
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 74 | 79
participants | 4 | 4

10. Other Pre Specified Outcome: Medical Outcomes Study (MOS) Sleep Scale Score
Description: Participant-rated questionnaire to assess sleep quality and quantity. Consists of 12-item questionnaires answered on a range of 1 to 6 for questions (Q) 3 to 12, 1 to 5 for Q1(some questions are reversed so that high score reflects more of the attributes); and Q2 answered on 0 to 24. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range multiplied by 100); total score range:0 to 100; higher score = greater intensity of attribute. The items contribute to each scale and are averaged to create 7 scale scores and 2 sleep scale index. Scales with at least one item answered was used to generate a scale score. Scales include; sleep disturbance (SD), sleep quantity, snoring, awaken short of breath (ASoB), somnolence, sleep adequacy and optimal sleep; and a 9-item overall sleep problems index(SPI) I and II Subscales range from 0-100 except for sleep quantity (SQ) ranging from0 to 24. Except for sleep quantity, higher scores=greater impairment.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 7, 14, 21 of stable dosing phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
units on a scale
  Baseline: SD (n=78,79) | 20.48 (18.869) | 22.26 (20.420)
  Baseline: Somnolence (n=78,79) | 64.70 (24.409) | 66.50 (24.529)
  Baseline: Adequacy (n=78,79) | 34.62 (27.666) | 34.18 (26.967)
  Baseline: Snore (n=78,79) | 26.67 (31.196) | 22.53 (30.444)
  Baseline: ASoB (n=78,79) | 14.10 (23.043) | 13.92 (23.173)
  Baseline: SQ (n=78,79) | 7.24 (1.505) | 7.18 (1.607)
  Baseline: Optimal sleep (n=78,79) | 0.58 (0.497) | 0.51 (0.503)
  Baseline: SPI I (n=78,79) | 40.85 (17.576) | 42.53 (15.314)
  Baseline: SPI II (n=78,79) | 41.04 (16.508) | 42.24 (14.486)
  Day 5 (TP): SD (n=67,78) | 22.46 (20.818) | 19.15 (21.942)
  Day 5 (TP): Somnolence (n=67,78) | 55.42 (27.834) | 58.89 (26.240)
  Day 5 (TP): Adequacy (n=67,78) | 35.82 (28.292) | 36.92 (27.648)
  Day 5 (TP): Snore (n=67,78) | 22.99 (29.182) | 18.46 (28.425)
  Day 5 (TP): ASoB (n=67,78) | 8.66 (15.657) | 11.54 (20.263)
  Day 5 (TP): SQ (n=67,78) | 7.04 (1.408) | 6.88 (1.494)
  Day 5 (TP): Optimal sleep (n=67,78) | 0.48 (0.503) | 0.55 (0.501)
  Day 5 (TP): SPI I (n=67,78) | 38.91 (17.315) | 38.46 (16.158)
  Day 5 (TP): SPI II (n=67,78) | 38.38 (17.252) | 38.14 (15.509)
  Day 10 (TP): SD (n=69,76) | 21.43 (20.637) | 16.94 (18.685)
  Day 10 (TP): Somnolence (69,76) | 58.55 (26.516) | 59.74 (25.979)
  Day 10 (TP): Adequacy (n=69,76) | 33.33 (27.422) | 35.66 (28.064)
  Day 10 (TP): Snore (n=69,76) | 19.71 (26.007) | 20.26 (27.999)
  Day 10 (TP): ASoB (n=69,76) | 12.17 (21.204) | 7.89 (15.690)
  Day 10 (TP): SQ (n=69,76) | 7.12 (1.255) | 6.99 (1.322)
  Day 10 (TP): Optimal sleep (n=69,76) | 0.58 (0.497) | 0.58 (0.497)
  Day 10 (TP): SPI I (n=69,76) | 40.10 (16.626) | 37.76 (15.929)
  Day 10 (TP): SPI II (n=69,76) | 39.70 (16.628) | 37.03 (14.711)
  Day 15 (TP): SD (n=67,74) | 22.03 (21.177) | 17.11 (20.585)
  Day 15 (TP): Somnolence (67,74) | 53.93 (26.072) | 58.11 (28.467)
  Day 15 (TP): Adequacy (n=67,74) | 36.27 (29.379) | 38.78 (29.188)
  Day 15 (TP): Snore (n=67,74) | 19.70 (26.627) | 16.49 (26.350)
  Day 15 (TP): ASoB (n=67,74) | 12.24 (22.551) | 11.35 (22.715)
  Day 15 (TP): SQ (n=67,74) | 6.90 (1.293) | 7.15 (1.279)
  Day 15 (TP): Optimal sleep (n=67,74) | 0.60 (0.494) | 0.64 (0.485)
  Day 15 (TP): SPI I (n=67,74) | 38.71 (18.294) | 36.67 (16.889)
  Day 15 (TP): SPI II (n=67,74) | 38.05 (17.748) | 36.28 (16.884)
  Day 20 (TP): SD (n=59,65) | 22.99 (21.611) | 16.46 (17.522)
  Day 20 (TP): Somnolence (59,65) | 56.05 (28.070) | 57.23 (28.720)
  Day 20 (TP): Adequacy (n=59,65) | 36.95 (28.723) | 43.85 (30.088)
  Day 20 (TP): Snore (n=59,65) | 22.37 (30.869) | 15.69 (23.316)
  Day 20 (TP): ASoB (n=59,65) | 10.85 (17.936) | 8.92 (20.625)
  Day 20 (TP): SQ (n=59,65) | 7.27 (1.257) | 7.40 (1.285)
  Day 20 (TP): Optimal sleep (n=59,65) | 0.69 (0.464) | 0.68 (0.471)
  Day 20 (TP): SPI I (n=59,65) | 39.32 (19.206) | 34.05 (16.240)
  Day 20 (TP): SPI II (n=59,65) | 38.65 (18.858) | 34.02 (16.200)
  Day 7 (SP): SD (n=63,67) | 20.73 (20.529) | 14.70 (18.250)
  Day 7 (SP): Somnolence (63,67) | 49.84 (29.883) | 57.81 (30.003)
  Day 7 (SP): Adequacy (n=63,67) | 40.63 (30.894) | 41.04 (29.032)
  Day 7 (SP): Snore (n=63,67) | 19.37 (29.614) | 20.90 (28.801)
  Day 7 (SP): ASoB (n=63,67) | 13.65 (23.231) | 8.96 (18.516)
  Day 7 (SP): SQ (n=63,67) | 7.05 (1.184) | 7.21 (1.297)
  Day 7 (SP): Optimal sleep (n=63,67) | 0.65 (0.481) | 0.66 (0.478)
  Day 7 (SP): SPI I (n=63,67) | 36.19 (18.597) | 34.98 (16.518)
  Day 7 (SP): SPI II (n=63,67) | 35.74 (18.159) | 34.43 (16.710)
  Day 14 (SP): SD (n=63,67) | 23.37 (22.364) | 16.55 (19.925)
  Day 14 (SP): Somnolence (63,67) | 51.53 (30.578) | 56.62 (28.554)
  Day 14 (SP): Adequacy (n=63,67) | 41.27 (32.353) | 42.09 (33.099)
  Day 14 (SP): Snore (n=63,67) | 19.37 (28.953) | 19.10 (27.509)
  Day 14 (SP): ASoB (n=63,67) | 12.38 (20.138) | 10.45 (19.183)
  Day 14 (SP): SQ (n=63,67) | 6.97 (1.282) | 7.19 (1.395)
  Day 14 (SP): Optimal sleep (n=63,67) | 0.63 (0.485) | 0.67 (0.473)
  Day 14 (SP): SPI I (n=63,67) | 37.99 (20.130) | 34.92 (19.283)
  Day 14 (SP): SPI II (n=63,67) | 37.27 (20.493) | 34.92 (18.611)
  Day 21 (SP): SD (n=56,61) | 21.27 (21.830) | 16.45 (17.791)
  Day 21 (SP): Somnolence (n=56,61) | 53.93 (30.252) | 55.08 (30.133)
  Day 21 (SP): Adequacy (n=56,61) | 35.71 (31.729) | 39.67 (30.874)
  Day 21 (SP): Snore (n=56,61) | 20.36 (29.168) | 20.98 (29.081)
  Day 21 (SP): ASoB (n=56,61) | 10.71 (17.874) | 6.89 (15.442)
  Day 21 (SP): SQ (n=56,61) | 6.95 (1.432) | 7.38 (1.227)
  Day 21 (SP): Optimal sleep (n=56,61) | 0.64 (0.483) | 0.69 (0.467)
  Day 21 (SP): SPI I (n=56,61) | 38.93 (19.354) | 35.52 (17.919)
  Day 21 (SP): SPI II (n=56,61) | 37.91 (19.436) | 34.78 (17.597)

11. Other Pre Specified Outcome: Number of Participants With Response to Sheehan Suicidality Tracking Scale (STS)
Description: Sheehan-STS is an 8-item clinician/participant administered prospective rating scale and an indicator of trigger assessment that tracks both treatment-emergent suicidal ideation and behaviors). Items 1a, 2-6, 8 scored on 5-point Likert scale (0=not at all, 1=a little, 2=moderately, 3=very, and 4=extremely). Items 1, 1b, 7, an indicator of trigger assessment (TA) require yes/no response. Items included 1= Ever suffer any accident, 1a= Extent plan/intend to hurt yourself, 1b= Intend to die, 2= Wish dead, 3= Want to harm yourself, 4= Think about suicide, 5= Plan for a suicide, 6= Prepare for suicide (PS) with intent to die (ITD), 7= Injure yourself on purpose, 8= Attempt suicide. Result for item 1 indicates if any of the participant ever suffered any accident, 1b indicates if any of the participant intended to die, 7 indicates if any of the participant injured themselves purposely and trigger assessment indicates if any of the participant evoked trigger assessment.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 7, 14, 21 of stable dosing phase
Population: FAS. Here "n" signifies participants who were evaluable at specified time points for each arm, respectively. Results for a parameter are not reported at certain time points since none of the participants were evaluable for the parameter at those time points.
Measure: Number; unit: participants
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
participants
  Baseline:Ever suffer any accident (n=78, 79) | 0 | 1
  Baseline:Hurt Yourself:Not at all (n=0,1) | 0 | 1
  Baseline:Wish dead:Not at all (n=78,79) | 77 | 79
  Baseline:Wish dead:A little (n=78,79) | 1 | 0
  Baseline:Harm yourself:Not at all (n=78,79) | 77 | 79
  Baseline:Harm yourself:A little (n=78,79) | 1 | 0
  Baseline:Think about suicide:Not at all (n=78,79) | 77 | 79
  Baseline:Think about suicide:A little (n=78, 79) | 1 | 0
  Baseline:Plan suicide:Not at all (n=78, 79) | 78 | 79
  Baseline:PS with ITD:Not at all (n=78, 79) | 78 | 79
  Baseline:Injure yourself on purpose (n=78,79) | 0 | 0
  Baseline:Attempt suicide:Not at all (n=78, 79) | 78 | 79
  Baseline:Trigger assessment (n=78, 79) | 1 | 0
  Day 5(TP):Ever suffer any accident (n=78,79) | 0 | 0
  Day 5(TP):Wish dead:Not at all (n=68,78) | 68 | 77
  Day 5(TP):Wish dead:A little (n=68, 78) | 0 | 1
  Day 5(TP):Harm yourself:Not at all (n=68,78) | 68 | 78
  Day 5(TP):Think about suicide:Not at all (n=68,78) | 68 | 78
  Day 5(TP):Plan suicide:Not at all (n=68,78) | 68 | 78
  Day 5(TP):PS with ITD:Not at all (n=68, 78) | 68 | 78
  Day 5(TP):Injure yourself on purpose (n=68,78) | 0 | 0
  Day 5(TP):Attempt suicide:Not at all (n=68,78) | 68 | 78
  Day 5(TP):Trigger assessment (n=68, 78) | 0 | 0
  Day 10(TP):Ever suffer any accident (n=69,76) | 0 | 0
  Day 10(TP):Intend to die (n=1,0) | 0 | 0
  Day 10(TP):Wish dead:Not at all (n=69, 76) | 69 | 76
  Day 10(TP):Harm yourself:Not at all (n=69,76) | 69 | 76
  Day 10(TP):Think About Suicide:Not at all(n=69,76) | 69 | 76
  Day 10(TP):Plan suicide:Not at all (n=69, 76) | 69 | 76
  Day 10(TP):PS with ITD:Not at all (n=69, 76) | 69 | 76
  Day 10(TP):Injure yourself on purpose (n=69,76) | 0 | 0
  Day 10(TP):Attempt suicide:Not at all (n=69, 76) | 69 | 76
  Day 10(TP):Trigger assessment (n=69, 76) | 0 | 0
  Day 15(TP):Ever suffer any accident (n=67,74) | 0 | 1
  Day 15(TP):Hurt Yourself:Not at all (n=0, 1) | 0 | 1
  Day 15(TP):Intend to die (n=2,0) | 0 | 0
  Day 15(TP):Wish dead:Not at all (n=67,74) | 67 | 74
  Day 15(TP):Harm yourself:Not at all (n=67,74) | 67 | 74
  Day 15(TP):Think about suicide:Not at all(n=67,74) | 67 | 73
  Day 15(TP):Think about suicide:A little (n=67,74) | 0 | 1
  Day 15(TP):Plan suicide:Not at all (n=67,74) | 67 | 74
  Day 15(TP):PS with ITD:Not at all (n=67,73) | 67 | 73
  Day 15(TP):Injure yourself on purpose (n=67,74) | 0 | 0
  Day 15(TP):Attempt suicide:Not at all (n=67, 74) | 67 | 74
  Day 15(TP):Trigger assessment (n=67,74) | 0 | 0
  Day 20(TP):Ever suffer any accident (n=58,64) | 0 | 0
  Day 20(TP):Wish dead:Not at all (n=58,64) | 58 | 63
  Day 20(TP):Wish dead:A little (n=58,64) | 0 | 1
  Day 20(TP):Harm yourself:Not at all (n=58,64) | 58 | 64
  Day 20(TP):Think about suicide:Not at all(n=58,64) | 58 | 64
  Day 20(TP):Plan suicide:Not at all (n=58,64) | 58 | 64
  Day 20(TP):PS with ITD:Not at all (n=58,64) | 58 | 64
  Day 20(TP):Injure yourself on purpose (n=58,64) | 0 | 0
  Day 20(TP):Attempt suicide:Not at all (n=58, 64) | 58 | 64
  Day 20(TP):Trigger assessment (n=58, 64) | 0 | 0
  Day 7(SP):Ever suffer any accident (n=63,67) | 0 | 0
  Day 7(SP):Intend to die (n=0,1) | 0 | 0
  Day 7(SP):Wish dead:Not at all (n=63,67) | 63 | 67
  Day 7(SP):Harm yourself:Not at all (n=63,67) | 63 | 67
  Day 7(SP):Think about suicide:Not at all(n=63,67) | 63 | 67
  Day 7(SP):Plan suicide:Not at all (n=63,67) | 63 | 67
  Day 7(SP):PS with ITD:Not at all (n=63,67) | 63 | 67
  Day 7(SP):Injure yourself on purpose (n=63,67) | 0 | 0
  Day 7(SP):Attempt suicide:Not at all (n=63,67) | 63 | 67
  Day 7(SP):Trigger assessment (n=63, 67) | 0 | 0
  Day 14(SP):Ever suffer any accident (n=63,67) | 0 | 0
  Day 14(SP):Intend to die (n=1,0) | 0 | 0
  Day 14(SP):Wish dead:Not at all (n=63,67) | 62 | 67
  Day 14(SP):Wish dead:A little (n=63,67) | 1 | 0
  Day 14(SP):Harm yourself:Not at all (n=63,67) | 63 | 67
  Day 14(SP):Think about suicide:Not at all(n=63,67) | 63 | 67
  Day 14(SP):Plan suicide:Not at all (n=63,67) | 63 | 67
  Day 14(SP):PS with ITD:Not at all (n=63, 67) | 63 | 67
  Day 14(SP):Injure yourself on purpose (n=63,67) | 0 | 0
  Day 14(SP):Attempt suicide:Not at all (n=63, 67) | 63 | 67
  Day 14(SP):Trigger assessment (n=64,67) | 0 | 0
  Day 21(SP):Ever suffer any accident (n=56, 61) | 0 | 0
  Day 21(SP):Wish dead:Not at all (n=56,61) | 56 | 61
  Day 21(SP):Harm yourself:Not at all (n=56,61) | 56 | 61
  Day 21(SP):Think about suicide:Not at all(n=56,61) | 56 | 61
  Day 21(SP):Plan suicide:Not at all (n=56,61) | 56 | 61
  Day 21(SP):PS with ITD:Not at all (n=56,61) | 56 | 61
  Day 21(SP):Injure yourself on purpose (n=56,61) | 0 | 0
  Day 21(SP):Attempt suicide:Not at all (n=56,61) | 56 | 61
  Day 21(SP):Trigger assessment (n=56,61) | 0 | 0

12. Secondary Outcome: Computer Based Objective Cognition Testing (CogState) Groton Maze Learning Task (GMLT)
Description: GMLT: a cognitive test which assessed executive function. Participant was shown a 10 multiplied by 10 grid of tiles on a computer touch screen. A 28-step pathway was hidden among 100 possible locations. The participant was instructed to move 1 step from the start location and then continue 1 tile at a time, toward the end to find the pathway. The outcome measure was total number of errors made in attempting to learn the same hidden pathway on 5 consecutive trials at a single session. Score ranges from 0 to infinity. Lower scores meant a better performance.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 21 of stable dosing phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
errors
  Baseline: n=78, 79 | 48.71 (19.91) | 53.19 (27.33)
  Day 5 (TP): n=72, 79 | 48.49 (21.24) | 48.32 (23.68)
  Day 10 (TP): n=72, 78 | 44.88 (15.41) | 43.59 (17.24)
  Day 15 (TP): n=67, 75 | 44.54 (16.73) | 44.36 (18.11)
  Day 20 (TP): n=60, 66 | 43.17 (17.09) | 45.47 (19.82)
  Day 21 (SP): n=61, 65 | 44.48 (17.45) | 47.02 (25.52)

13. Secondary Outcome: Computer Based Objective Cognition Testing (CogState) Detection Speed
Description: Detection speed: a cognitive test which assessed psychomotor function. A playing card was presented face up in the center of the screen. As soon as this happened, the participant was to press the 'Yes' key. The outcome measure was speed of performance; mean of the log10 transformed reaction time for correct responses [measured in log10 milliseconds (msec)]. Scores ranges from 2 (best) to 3.3 (worst). Lower scores meant a better performance.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 21 of stable dosing phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 msec
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
log10 msec
  Baseline: n=78, 79 | 2.55 (0.13) | 2.55 (0.12)
  Day 5 (TP): n=73, 79 | 2.51 (0.1) | 2.52 (0.11)
  Day 10 (TP): n=72, 78 | 2.52 (0.1) | 2.52 (0.1)
  Day 15 (TP): n=67, 75 | 2.53 (0.12) | 2.53 (0.1)
  Day 20 (TP): n=60, 66 | 2.52 (0.11) | 2.52 (0.11)
  Day 21 (SP): n=61, 64 | 2.54 (0.12) | 2.54 (0.1)

14. Secondary Outcome: Computer Based Objective Cognition Testing (CogState) Identification Speed
Description: Identification speed: a cognitive test which assessed visual attention. A playing card was presented face up in the center of the screen. As soon as this happened, the participant had to decide whether the card was red or not. The outcome measure was speed of performance; mean of the log10 transformed reaction time for correct responses (measured in log10 msec). Score ranges from 2 (best) to 3.3 (worst). Lower scores meant a better performance.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 21 of stable dosing phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 msec
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 78 | 79
log10 msec
  Baseline: n=78, 79 | 2.74 (0.11) | 2.72 (0.10)
  Day 5 (TP): n=72, 79 | 2.72 (0.09) | 2.72 (0.09)
  Day 10 (TP): n=72, 78 | 2.72 (0.10) | 2.73 (0.10)
  Day 15 (TP): n=67, 75 | 2.73 (0.09) | 2.73 (0.09)
  Day 20 (TP): n=60, 66 | 2.72 (0.08) | 2.73 (0.11)
  Day 21 (SP): n=61, 65 | 2.73 (0.10) | 2.73 (0.10)

15. Secondary Outcome: Computer Based Objective Cognition Testing (CogState) One Card Learning
Description: One card learning: a cognitive test which assessed visual learning. Participants were to remember which cards were previously shown in a task. The outcome measure was accuracy of performance; arcsine transformation of the square root of the proportion of correct responses. Score ranges from 0 (worse) to 1.57 (best). Higher scores meant a better performance.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 21 of stable dosing phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: arcsine (square root proportion correct)
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 77 | 79
arcsine (square root proportion correct)
  Baseline: n=77, 79 | 1.01 (0.15) | 1.02 (0.13)
  Day 5 (TP): n=72, 79 | 1.01 (0.14) | 1.02 (0.13)
  Day 10 (TP): n=72,78 | 1.01 (0.13) | 1.02 (0.12)
  Day 15 (TP): n=67, 75 | 1.00 (0.14) | 1.01 (0.14)
  Day 20 (TP): n=59, 66 | 1.02 (0.17) | 1.02 (0.17)
  Day 21 (SP): n=61, 65 | 1.01 (0.16) | 1.02 (0.16)

16. Secondary Outcome: Computer Based Objective Cognition Testing (CogState) Continuous Paired Associate Learning (CPAL)
Description: CPAL: a cognitive test which assessed visual episodic learning. Participant was to learn and remember picture locations on the screen and was to tap the target on the central location to begin. As each picture was revealed, the participant was to remember where the picture was located and tap that location. The outcome measure was the number of errors made in correctly placing each of the 4 patterns in their location 4 times. Score ranges from 0 to infinity. Lower scores meant a better performance.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 21 of stable dosing phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 74 | 78
errors
  Baseline: n=74, 75 | 48.42 (57.11) | 46.4 (52.59)
  Day 5 (TP): n=71, 77 | 37.18 (48.03) | 37.01 (48.86)
  Day 10 (TP): n=70, 78 | 36.64 (54.25) | 30.54 (42.4)
  Day 15 (TP): n=66, 75 | 27.59 (36.84) | 25.52 (37.39)
  Day 20 (TP): n=59, 65 | 29.9 (40.17) | 19.49 (27.69)
  Day 21 (SP): n=61, 64 | 31.75 (42.8) | 24.98 (32.13)

17. Secondary Outcome: Computer Based Objective Cognition Testing (CogState ) Composite Score
Description: CogState had 5 outcome measures that measured the cognitive constructs. GMLT, detection, identification, one card learning and CPAL. GMLT score range: 0 (best) to infinity (worst), detection and identification score range: 2 (best) to 3.3 (worst); One card learning score range: 0 (worse) to 1.57 (best) and CPAL score range: 0 (best) to infinity (worst). The individual score was standardized at each assessment and was then averaged to yield a composite score; total possible score: minus infinity to plus infinity. Positive composite score=improved performance.
Time Frame: Baseline, Day 5, 10, 15, 20 of titration phase; Day 21 of stable dosing phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-03654746 | Placebo
Number analyzed (Participants) | 74 | 79
Units on a scale
  Baseline: n=74, 79 | 0.02 (0.72) | 0.06 (0.6)
  Day 5 (TP): n=73, 79 | 0.19 (0.62) | 0.19 (0.58)
  Day 10 (TP): n=72, 78 | 0.21 (0.58) | 0.23 (0.55)
  Day 15 (TP): n=67, 75 | 0.19 (0.54) | 0.21 (0.53)
  Day 20 (TP): n=60, 66 | 0.24 (0.56) | 0.25 (0.59)
  Day 21 (SP): n=61, 65 | 0.16 (0.67) | 0.17 (0.66)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-03654746 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/78 | 1/79
Other Adverse Events (participants affected / at risk) | 48/78 | 43/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03654746 (N=78) | Placebo (N=79)
Injury (Injury, poisoning and procedural complications) | 1 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03654746 (N=78) | Placebo (N=79)
Palpitations (Cardiac disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Eye irritation (Eye disorders) | 1 | 1
Eye swelling (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 6
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 3
Chest pain (General disorders) | 2 | 1
Fatigue (General disorders) | 0 | 1
Feeling cold (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Feeling jittery (General disorders) | 0 | 1
Irritability (General disorders) | 3 | 1
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Swelling (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5
Otitis externa (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Semen volume decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 10 | 6
Migraine (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 1
Abnormal dreams (Psychiatric disorders) | 2 | 0
Aggression (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 8 | 3
Middle insomnia (Psychiatric disorders) | 2 | 2
Mood altered (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Nicotine dependence (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 2 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Tension (Psychiatric disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.